CLINICAL TRIAL: NCT07382167
Title: A 26-Week, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Tenapanor for the Treatment of Chronic Idiopathic Constipation (CIC) in Adults
Brief Title: A 26-Wk Study to Assess Safety & Efficacy of Tenapanor for T/t of Chronic Idiopathic Constipation in Adults
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEN-03-301
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Idiopathic Constipation (CIC)
Keywords: CIC
MeSH Terms: interventions — tenapanor; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tenapanor 5 mg BID (Experimental): Patients will be randomized to receive 5 mg tenapanor twice daily.
  Interventions: Drug: Tenapanor 5 mg BID
- Tenapanor 25 mg BID (Experimental): Patients will be randomized to receive 25 mg tenapanor twice daily.
  Interventions: Drug: Tenapanor 25 mg BID
- Tenapanor 50 mg BID (Experimental): Patients will be randomized to receive 50 mg tenapanor twice daily.
  Interventions: Drug: Tenapanor 50 mg BID
- Placebo Comparator (Placebo Comparator): Patients will be randomized to receive matching placebo twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor 5 mg BID — Patients will receive tenapanor 5 mg BID (total of 10 mg daily)
  Arms: Tenapanor 5 mg BID
Drug: Tenapanor 25 mg BID — Patients will receive tenapanor 25 mg BID (total of 50 mg daily)
  Arms: Tenapanor 25 mg BID
Drug: Tenapanor 50 mg BID — Patients will receive tenapanor 50 mg BID (total of 100 mg daily)
  Arms: Tenapanor 50 mg BID
Drug: Placebo — Patients will receive matching placebo BID
  Arms: Placebo Comparator

SUMMARY:
This is a 26-week, multi-center, randomized, double-blind, placebo-controlled study with a 4-week treatment-free Safety Follow-up period to assess the safety and efficacy of tenapanor (5 mg, 25mg, and 50 mg) in adult patients with Chronic Idiopathic Constipation (CIC) when administered twice daily for 26 consecutive weeks.

DETAILED DESCRIPTION:
This study consists of a 2-week Screening period, followed by a 26-week randomized treatment period (RTP), and a 4-week treatment-free Safety Follow-up period.

After obtaining study informed consent from patients, the 2-week Screening period starts. Patients will be fully assessed for eligibility into the study. The assessments will include evaluation of inclusion/exclusion criteria, including medical histories, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests.

Patients will also self-report, on information about the status of their constipation symptoms and severity via an electronic diary (eDiary). Patient compliance with the eDiary will be monitored to determine eligibility at the end of screening.

Eligible patients will be randomized (Visit 2) to receive tenapanor 5 mg BID, 25 mg BID, 50 mg BID, or placebo for 26 consecutive weeks as the double-blind RTP. During this period, patients will continue recording daily assessments of constipation symptoms and weekly assessments of constipation severity in the eDiary. Patients will have return visits every two to six weeks at Weeks 2, 4, 8, 12, 16, 20 and 26(Visit 3-9) to undergo safety assessments.

Upon completion of the 26-week RTP, patients will be monitored for AEs during the 4-week treatment-free Safety Follow-up period and complete the Follow-up visit (Visit 10) at the end of this period to undergo safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that are ≥18 to ≤80 years old at the Screening visit (Visit 1).
2. Meet the Rome IV Diagnostic Criteria for functional constipation.
3. Females of non-childbearing potential, or agree to the use of an acceptable means of contraception for up to 30 days following the last dose of study medication.
4. Males must agree to use an appropriate method of barrier contraception (e.g., latex condom with a spermicidal agent) or have documented surgical sterilization.
5. Meets the entry criteria assessed during the Screening period.
6. Ability to understand and provide input on the assessments in the eDiary.
7. Provide written informed consent before the initiation of any study-specific procedures.
8. Must agree to have daily access to eDiary via a computer, tablet or smart phone

Exclusion Criteria:

1. Loose or watery stool (BSFS of 6 or 7) in the absence of any medication that is known to affect stool consistency (i.e., prohibited medicine) for >25% of bowel movements (BMs) during the 3 months prior to the Screening visit
2. Fecal impaction within 6 months prior to the Screening visit
3. Unexplained and clinically significant "alarm symptoms" including lower gastrointestinal (GI) bleeding, iron-deficiency anemia, weight loss or fever of unknown origin
4. Functional diarrhea as defined by Rome IV criteria
5. IBS with constipation (IBS-C), IBS with diarrhea (IBS-D), mixed IBS (IBS-M), or unsubtyped IBS as defined by Rome IV criteria
6. Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract within 6 months prior to the Screening visit, or active disease within 6 months prior to the Screening visit
7. Patient with central nervous system disorder (e.g., Parkinson's disease, spinal cord injury, or multiple sclerosis)
8. Use of prohibited medications defined by protocol
9. Patient has a history or current evidence of laxative abuse
10. Hepatic dysfunction (ALT [SGPT] or AST [SGOT] >2.5 times the upper limit of normal) or renal impairment (serum creatinine >2 mg/dL)
11. Positive HIV, hepatitis B or hepatitis C test at screening
12. Positive urinary drug test at Screening, with the exception of cannabis and cannabidiol (CBD)
13. Any evidence of or treatment of malignancy within 1 year prior to the Screening visit
14. Any surgery on the stomach, small intestine or colon; appendectomy or cholecystectomy are not excluded unless within 60 days prior to the Screening visit
15. Pregnant women or women planning to become pregnant during trial participation
16. A major psychiatric disorder (DSM-III-R or DSM-IV) including major depression or other psychoses that has required hospitalization in the last year prior to the Screening visit.
17. Alcohol or substance abuse within 1 year prior to the Screening visit
18. Participation in other clinical trials within 1 month prior to the Screening visit
19. Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, neurologic, psychiatric or any disease that may interfere with the patient's successful completion of the trial
20. Patient is involved in the conduct and/or administration of this trial as an Investigator, Sub-Investigator or other staff member, or is a first-degree family member or relative residing with one of the above persons involved in the trial
21. If, in the opinion of the Investigator, the patient is unable or unwilling to fulfill the requirements of the protocol or has a condition, which would render the results uninterpretable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Durable CSBM response | 12 Weeks
  Durable CSBM response is defined as achieving the weekly CSBM response for ≥9 out of the first 12 weeks of the RTP and and for ≥3 of the last 4 weeks of the first 12 weeks of RTP

SECONDARY OUTCOMES:
9/12 week CSBM response | 12 Weeks
  9/12 week CSBM response defined as achieving the weekly CSBM response for ≥9 out of the first 12 weeks of the RTP
Change from baseline in CSBM frequency | 12 Weeks
  Change from baseline over the first 12 weeks of the RTP in CSBM frequency
Change from baseline in SBM frequency | 12 Weeks
  Change from baseline over the first 12 weeks of the RTP in SBM frequency
Change from baseline in stool consistency | 12 Weeks
  Change from baseline over the first 12 weeks of the RTP in stool consistency
Change from baseline in stool straining | 12 Weeks
  Change from baseline over the first 12 weeks of the RTP in straining

CONTACTS AND LOCATIONS:
Overall Officials: Susan Edelstein, PhD, Study Director — Ardelyx Inc
Locations (32):
- United States (32):
  - Elite Clinical Studies, Phoenix, Arizona
  - Arkansas Gastroenterology - North Little Rock, North Little Rock, Arkansas
  - Erick H. Alayo Medical Corporation, Chula Vista, California
  - Proactive Clinical Research, Fort Lauderdale, Florida
  - Suncoast Clinical Research, Inc. - New Port Richey, New Port Richey, Florida
  - DelRicht Clinical Research - Atlanta, Atlanta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - DelRicht Clinical Research - Indianapolis, Indianapolis, Indiana
  - DelRicht Clinical Research - Overland Park, Overland Park, Kansas
  - DelRicht Clinical Research - Louisville, Louisville, Kentucky
  - DelRicht Clinical Research - Covington, Mandeville, Louisiana
  - DelRicht Clinical Research - New Orleans, New Orleans, Louisiana
  - DelRicht Clinical Research - Prairieville, Prairieville, Louisiana
  - DelRicht Clinical Research - Gulfport, Gulfport, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - DelRicht Clinical Research - Town and Country, Town and Country, Missouri
  - Excel Clinical Research, Las Vegas, Nevada
  - Advanced Research Institute - Reno, Reno, Nevada
  - Albuquerque Clinical Trials (ACT), Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Peters Medical Research, High Point, North Carolina
  - Lucas Research - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Remington Davis, Inc., Columbus, Ohio
  - Advanced Research Institute - Portland, Tigard, Oregon
  - DelRicht Clinical Research - Charleston, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Zenos Clinical Research, Dallas, Texas
  - EPIC Medical Research, DeSoto, Texas
  - North Hills Medical Research Inc. (North Hills Family Medicine), North Richland Hills, Texas
  - DelRicht Clinical Research - McKinney, Prosper, Texas
  - Advanced Research Institute - Ogden, Ogden, Utah
  - Advanced Research Institute - Sandy, Sandy City, Utah

IPD SHARING:
Plan to Share IPD: No